CLINICAL TRIAL: NCT05438433
Title: Outcome of Preservation of Mitral Valve Leaflets During Mitral Replacement
Brief Title: Outcome of Preserved Mitral Valve Apparatus During Mitral Valve Replacement
Acronym: EarlyOutcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Hamdy Dosoky Ibraheem Elayouty, Prof. of Cardio-thoracic Surgery, Suez Canal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2796#
Record Dates: First submitted 2022-06-01; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Diseases of Mitral Valves; Abnormality of Mitral Valve Annulus (Disorder); Mitral Valve Replacement
Keywords: : Preservation of mitral apparatus ,; mitral valve replacement; Rheumatic valve disease and ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: both groups of patients received surgical treatment parallel to each other.
Masking Description: All roles were unmasked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Sham Comparator): 50 patients with isolated rheumatic mitral valve disease (group A)
  Interventions: Device: St.Jude bi leaflet prosthetic mitral valve to replace the diseased valve with preservation of both leaflets
- Group B (Other): 50 patients with mitral disease and myocardial ischemia (group B)
  Interventions: Device: St.Jude bi leaflet prosthetic mitral valve to replace the diseased valve with preservation of both leaflets

INTERVENTIONS:
Device: St.Jude bi leaflet prosthetic mitral valve to replace the diseased valve with preservation of both leaflets — St.Jude prosthetic(FDA approved) mitral valve replacement with or without coronary artery bypass grafts
  Other Names: St.Jude bi leaflet prosthesis to replace diseased valve with preservation of leaflets with Myocardial re-vascularization; St.Jude prosthetic mitral replacement with preservation of valve apparatus and bypass grafts for associated coronary artery disease

SUMMARY:
Are there differences in outcome of mitral valve replacement with preservation of mitral apparatus among rheumatic and/or ischemic mitral lesions?.

Mitral valve replacement with preservation of leaflets, and added coronary artery-bypass surgery, when indicated, is it a feasible and reproducible procedure?.

The study was designed to compare outcome after prosthetic mitral replacement with preservation of mitral apparatus for rheumatic valve disease with outcome of replacement for ischemic myocardium and mitral valve disease, The outcomes will be guided by clinical assessment. and echo-cardiograph.

DETAILED DESCRIPTION:
Objectives: The aim is to compare outcome of modified preservation of mitral valve apparatus during prosthetic mitral replacement for rheumatic versus myocardial ischemia &mitral valve disease.

Methods ;This prospective cross-sectional comparative study will include 50 patients with isolated rheumatic mitral valve disease (group A) and 50 patients with mitral disease and myocardial ischemia (group B), surgery is expected to be performed between 2017 and 2020 at one center. All patients will have modified preservation of mitral apparatus during prosthetic mitral replacement. Additionally, group B patients will have bypass grafts to left anterior descending and/or posterior descending / right coronary artery. Data will be collected and analyzed.

The Institutional Review Board (IRB), Ethics Committee (EC)-approval and consent of each patient were obtained.

Criteria for inclusion of patients and exclusion of others were determined according to the guide lines.

Statistical analysis::

Qualitative variables and their association among both groups were studied by applying Chi-square test and Fisher Exact test. Quantitative variables among both groups were compared by applying independent samples t-test. P < 0.05 values mean statistically-significant results.

ELIGIBILITY:
Inclusion Criteria::

Mitral stenosis (MS)

* symptoms are severely limiting and cannot be managed with diuresis and heart rate control.

Mitral regurgitation(MR):

* acute severe MR require surgical correction for hemo-dynamics and relief of symptoms .

Chronic primary mitral regurgitation:

* rheumatic heart disease: replacement before irreversible changes occur can be curative.

Mixed Mitral Stenosis and Mitral Regurgitation:

* If beta blockers and diuretics do not relieve symptoms, replacement should be performed only in patients who have severe limiting symptoms.
* Myocardial ischemia associating or complicated with miral valve disease.

Exclusion criteria

* Patients showing good response to medical therapy, and Cases complicated by:
* ineffective endocarditis,
* previous myocardial re-vascularization
* ischemic ventricular septal defect,
* left ventricular aneurysm,
* Ruptured papillary muscles of mitral apparatus.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Smoking index | One week before surgery(or during first clinical visit) .
  Number of Packs every day X number of years of smoking= Pack.year,
Age and gender for each participant | One week before surgery .
  Males above 40 years and Females above 45 years need pre-operative coronary angio-graph
For each participant: pathological:type of mitral valve lesion | Seven days before surgery .
  severe stenosis with mitral area < 1 cm square, severe regurgitation, or mixed lesions
For each participant: etiological :type of mitral valve lesion | Seven days before surgery .
  Rheumatic: distorted thickened leaflets,thickened fibrosed chordae
For each participant: etiological :type of mitral valve lesion | Seven days before surgery- echo-cardiograph.
  Rheumatic: distorted thickened leaflets,thickened fibrosed chordae or ischemic incompetence
For each participant:, assessing sub-valvular apparatus | One week before surgery. with Echo-cardiograph.
  Thickened chordae, ruptured chordae, ischemia of papillary muscles or lateral ventricular wall.
Abascal echo-cardiographic mitral valve score (Wilkins score) | One week before surgery.with Echo-cardiograph
  :if score is 8 or less it is good for balloon valvo-plasty, if > 8 surgery is recommended ( leaflet mobility, thickness and calcification. Fourthly, sub-valvular thickening., higher scores = more deterioration
left ventricular wall motion abnormality | one week before surgery - with an echo-cardiograph
  hypokinesia, Akinesia, Dyskinesia of certain segment(s)
Number of participants with Signs of left ventricular dysfunction | seven days before surgery echo-cardiograph examination
  low ejection fraction <52%, low stroke volume< 70 ml, low cardiac output <5 litres per minute
Number of participants with pre-operative coronary artery disease | seven days before surgery, coronary angio-graph
  Expected on clinical bases and .proved by Echo-cardiograph-findings
Number of participants with pre-operative ischemic complications | seven days before surgery echo-cardiograph examination
  left ventricular thrombi, septal and left ventricular wall thickness in mm .
Assessment of any evolving new prosthetic valve dysfunction | intra-operative trans-esophageal echo-cardiograph examination
  Left atrioventricular outflow stenosis, prosthetic dysfunction due to preservation of valve apparatus
Change in post-operative left ventricular functions | 5 days post-operatively and end of 6th and 12 months after surgery with Echo-Cardiograph
  : Low Fractional Shortening < 28% , Ejection fraction < 40%,, increased left ventricular dimensions and volume
Change of Prosthetic mitral valve functions | Monthly through study completion up to 12 months after surgery..... with Echo-cardiograph
  Development of para-valvular leak or central jet of regurgitation or stuck valve by a thrombus

SECONDARY OUTCOMES:
changes on Clinical examination | Monthly up to 12 months after surgery)
  local and general Examination,: a new murmur, evolving heart failure
Changes in Results of Prothrombin time, concentration and.International normalized ratio | .Monthly through study completion up to 12 months.
  Adjust dose of oral anticoagulant.( between double and half to three times the control) Dose usually ranges between 1 and 11 mg warfarin tablet daily.
Mortality and Morbidity | Monthly through study completion up to 12 months.
  cause of mortality, type of morbidity: wound infection, hypertrophied scar, Kiloid Formation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. allaban, PhD, Study Director — Suez Canal University, FOM- Research Ethics Committee
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All authors contributed to the study conception and design. Material preparation, data collection and analysis were performed by H. D. Elayouty, H. S. Hassan and S.A. Elhafeez. The first draft of the manuscript was written by A. H.Elayouty and all authors commented on previous versions of the manuscript. All authors read and approved the final manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 360 days
Access Criteria: h.dosoky@yahoo.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT05438433/Prot_SAP_000.pdf